CLINICAL TRIAL: NCT06208800
Title: Effects of Inhaled Blend Aromatherapy on Sleep Duration, Sleep Quality, Time to Fall Asleep and Cognitive Level in Elderly People
Brief Title: The Effect of Aromatherapy on Sleep and Cognitive Level in the Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, BELÇİM EDE SARIKAYA, Internal Medicine Nurse MSc, Lecturer, Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-95961207-604.01.01-3755
Record Dates: First submitted 2023-12-09; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Insomnia; Cognitive Impairment; Elderly
Keywords: Aromatherapy; Sleep; Cognitive Functions; Elderly; Insomnia; Peppermint; Palmarosa; Musk sage; Petitgrain; Vetiver; Cedrus; Citrus Paradisi
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group to which the essential oil mixture will be applied (Experimental): Thirty elderly individuals will be included in the experimental group. The elderly individuals in the intervention group were given essential oil mixtures in 5 ml bottles prepared by the expert aromatherapist and the researcher, and it was decided to inhale these essential oils by dropping 5 drops on cotton wool for 10 minutes each for 4 weeks.
  Interventions: Other: Blend Aromatherapy
- Experimental group without essential oil mixture.Control group (No Intervention): Thirty elderly individuals will be included in the control group. This group will not be intervened, only questionnaires will be administered.

INTERVENTIONS:
Other: Blend Aromatherapy — Inhalation of a mixture of essential oils of peppermint, palmarosa for 10 minutes at 11:00 am during the day and vetiver, cedar, clary sage, musk sage, grapefruit and petitgrain for 10 minutes at 21:30 pm before bedtime for 4 weeks
  Arms: Experimental group to which the essential oil mixture will be applied

SUMMARY:
This research aims to investigate the effect of aromatherapy on sleep duration, sleep quality, falling asleep time and cognitive functions of elderly individuals in the short term and to improve the general health status and quality of life of elderly individuals in the long term.

DETAILED DESCRIPTION:
Due to the aging of the world population, the elderly population is increasing and age-related physiological changes and a number of health problems arise. Aging brings challenges such as chronic diseases, balance disorders, osteoporosis, disorientation, sleep disorders, neurological and psychiatric disorders. Changes during the aging process affect individuals' sleep duration, quality and cognitive level. Insufficient and poor quality sleep can lead to depression, anxiety, pain sensitivity, irritability, suppression of the immune system, decreased mental activity, in short, deterioration of general health and functioning. Sleep problems and some cognitive functions can be treated with pharmacological and non-pharmacological methods, but pharmacological methods can cause serious side effects and complications. Aromatherapy is a complementary alternative treatment method used for the physical, mental and spiritual positive effects of plant-derived essential oils. In our literature review, it was observed that some non-pharmacological approaches (such as massage, listening to music, phototherapy, relaxation exercises and aromatherapy) applied to different populations improved sleep problems and cognitive levels. There are studies in the literature evaluating the effect of aromatherapy, especially aromatherapy applied through massage, on sleep in the elderly, but there is no study examining the effect of inhaled mixture aromatherapy on insomnia, sleep duration, sleep quality, and time to fall asleep. and the interoperation of cognitive functions. However, as mentioned above, sleep problems and daytime sleepiness affect cognitive functions. This research, which was planned to fill this gap in the literature, has a unique value that distinguishes it from other studies on the subject.

The main purpose of the research is to examine the effect of blended aromatherapy applied via inhalation to elderly individuals on sleep duration, sleep quality, time to fall asleep and cognitive functions. For this purpose, an application was made to the elderly care center affiliated with the Ministry of Family and Social Services for research permission. Permission was obtained from the institution to conduct the research. In order to conduct the research, informed consent forms will be obtained from elderly individuals living in the elderly care center who have the ability to understand and answer the questions and those who do not have any knowledge. Those who have a disability to participate in the applications and those who meet the inclusion criteria will be identified and their participation in the research will be ensured. The minimum number of participants planned to be reached in the research was determined as 60. First of all, the elderly individuals will be equally distributed as experimental and control groups by simple randomization method. Then, after the elderly individuals in both groups are informed about the study, the survey and forms will be applied and they will be given a wearable smart watch and an Android mobile phone compatible with this watch to wear on their wrists for 4 days. The researcher will make the elderly in the intervention group smell peppermint and palmarosa oils for 10 minutes at 11:00 during the day for 4 weeks. In addition, the researcher will make the elderly in the experimental group smell the essential oil mixture of vetiver, cedar, clary sage, grapefruit and petitgrain for 10 minutes at 21:30 in the evening before going to bed on the same day. Essential oil mixture inhalation will not be applied to the control group. The researcher planned to re-administer the questionnaires and forms to the experimental and control groups at the beginning of the application and at the end of the 4th week. It is planned to give individuals in both the experimental group and the control group a wearable smart watch worn on the wrist and an Android mobile phone compatible with the smart watch until the end of the 4th week. Thanks to the application on the Android mobile phone, the data from the smart watch will be transferred to the computer. The obtained values will be transferred to the Social Sciences Statistical Package (SPSS) 22.0 statistical analysis program and the necessary analyzes will be performed.

It is planned to provide materials and consumables in the first three months of the research, to obtain data in seven months, and to interpret the results with statistical analysis in the last two months. The data obtained as a result of the research will pave the way for the development of new strategies to improve the sleep quality and cognitive levels of elderly individuals. The research aims to investigate the effects of aromatherapy on the sleep duration, sleep quality, time to fall asleep and cognitive functions of elderly individuals in the short term. In the long term, it will contribute to improving the general health status of elderly individuals, increasing their quality of life and improving their general health status. This research, which is one of the rare studies in the literature, will shed light on future research in this field and has the power to appear as articles in important international journals and to be presented as papers at scientific meetings.

ELIGIBILITY:
Inclusion Criteria:

* 65 -85 years of age
* Not having a condition that prevents him/her from participating in the practices (such as pain, severe infection)
* Acceptance to participate in the research,
* Not having a psychiatric problem that prevents them from working and not being diagnosed with mental deficiency,
* To be capable of understanding and answering the questions,
* No hearing or speech impairment and no problem with smell that would hinder communication,
* Any respiratory system disease (such as asthma, COPD), allergic skin disease (such as eczema) and no history of allergy to plants,
* No known allergy to the essential oils to be used,
* At the time of the study, any of the traditional and complementary medicine practices is not using it,
* Daytime sleepiness (Epworth Sleepiness Scale Score ≥ 11),
* Pittsburgh Sleep Quality Index (PUKI) score ≥ 5

Exclusion Criteria:

* Antidepressants, antihistamines, diuretics, hypnotics, benzodiazepines that affect sleep quality and the use of narcotic analgesics,
* Body Mass Index (BMI) ≥ 30,
* 5 and above, expressing that he/she has pain,
* Allergy to any odor or plant,
* Presence of a respiratory disease such as asthma and chronic obstructive pulmonary disease

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-30 (Estimated); Primary Completion 2024-03-29 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Elderly Introduction Form | Four Weeks
  The Elderly Introduction Form is a form prepared by the researcher by scanning the literature and contains information about the sociodemographic characteristics of individuals (age, gender, BMI, chronic disease, etc.) (Her and Cho, 2021; Aydın Yıldırım and Kitiş, 2020).
Epworth Sleepiness Scale | Four Weeks
  It is a scale used to indicate daytime sleepiness and sleepiness tendency during the day. It consists of 8 questions in total. Each question is filled in by the individual himself, giving 0-3 points. In this survey, the individual's likelihood of falling asleep in certain situations on a normal day when he or she is not overly tired is questioned. The scoring method is the same for all questions; if there is no probability of falling asleep, 0 is given, if there is a low probability of falling asleep, 1, if there is a medium probability, 2 and if there is a high probability, 3 points are given. If the total score is between 0-10, it indicates normal condition for healthy individuals, between 11-14, it indicates mild sleepiness, between 15-17, it indicates moderate sleepiness, and if it is 18 and above, it indicates the presence of excessive daytime sleepiness.
Pittsburgh Sleep Quality Index-PSQI | Four Weeks
  PSQI , is a safe and consistent questionnaire that evaluates the amount of sleep, sleep quality, presence and severity of sleep disorder in individuals in the last month, and was adapted into Turkish by Ağargün by. PSQI consists of 12 questions in total. The evaluation score of an item is between 0-3. In this way, the total score obtained from all 7 components gives the total PSQI score. The total score obtained varies between 0-21. The higher the score, the worse the sleep quality. A score greater than five indicates poor sleep quality
Blessed Orientation Memory Concentration Test (BOBKT) | Four Weeks
  The test was developed by Blessed, Tomlinson and Roth in 1968 and consists of 26 items. The first and second questions are related to time orientation and ask for the current month and year. It is then made to memorize a memory item containing information (a fictitious first name, a surname, a fictitious street name, an imaginary number, and a fictitious city name). The fourth and fifth questions are questions designed to measure attention. In the fourth question, the patient is asked to count back from twenty, one by one. In the fifth question, it is expected that the person will count the months backwards. Then, the last question is the memory measurement question, in which the individual is asked about the memorized memory item. An increase in the score indicates a decrease in cognitive functions. This test, which has been standardized into Turkish, can be applied to individuals at all educational levels since it is not related to the year of education (Akça-Kalem et al., 2002).
Wearable Smart Device Worn on the Wrist | Four Weeks
  Wearable technologies, which have become very popular especially in the field of healthcare, monitor the health status of patients remotely and send the data to the physician without the need for outpatient clinic visits. In this way, unnecessary procedures are prevented, costs are reduced and the quality of health services is increased.These wearable smart devices are devices that allow continuous measurement every second. In this research, it is planned to objectively obtain individuals' falling asleep time, awake time, bedtime, wake-up time, REM sleep, light and deep sleep hours, snoring and total sleep time throughout the night, with a smart watch worn on the wrist It is planned to analyze these recorded data with a statistical program and to interpret and transfer them in detail in the findings section of the research.
Android Mobile Phone | Four Weeks
  They are Android devices that are compatible with the watch required for the operation of wrist-worn smart watches and the transfer of data from the smart watch.

CONTACTS AND LOCATIONS:
Overall Officials: Belçim EDE SARIKAYA, MSc, Principal Investigator — İstanbul Medipol University; Sebahat ATEŞ, PhD, Principal Investigator — Üsküdar University; Ayşe Arzu SAYIN ŞAKUL, PhD, Principal Investigator — İstanbul Medipol University; Tuğba KAMAN, PhD, Principal Investigator — Üsküdar University
Locations (1):
- İstanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No